CLINICAL TRIAL: NCT05013710
Title: Evaluating the Mobile Clinic Model as a Means of Increasing Access to Reproductive and Sexual Health
Acronym: MHCE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Plan A Health, Inc (Other)
Collaborators: Organon (Industry)
Responsible Party: Principal Investigator, Caroline Weinberg, Executive Director, Plan A Health, Inc
Other Study IDs: 01
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthcare Disparities; Reproductive Health; Sexual Health; Program Evaluation; Health Care Quality, Access, and Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Plan A Health: Founded in 2018, Plan A Health, Inc seeks to address health care disparities in rural communities by improving access to reproductive and sexual care. Beginning April 2021, the first Plan A mobile health clinic opened, serving five counties in the Mississippi Delta. The care team in the clinic includes a community health worker, nurse practitioner, volunteer providers, residents, and a collaborating physician.
  Interventions: Other: Complete Clinical Interaction
- Just the Pill: Just The Pill offers telemedicine appointments by phone or online for sexual and reproductive health needs that is delivered to the patient's home. The organization is also opening a mobile health clinic that will deliver care directly to communities.
  Interventions: Other: Complete Clinical Interaction
- University of Florida Mobile Outreach Clinic: The mission of the Mobile Outreach Clinic is to reduce health disparities by providing best practice, flexible, low-barrier primary care at no cost to patients unable to access the healthcare system. They focus on addressing the social barriers that drive health inequities and educating health professions students in an environment that equips them to become the socially conscious medical providers of the future.
  Interventions: Other: Complete Clinical Interaction

INTERVENTIONS:
Other: Complete Clinical Interaction — The intervention consists of a completed interaction with the mobile health clinic during the study periods, on which adequate evaluative data was collected on the patient visit (e.g. staff was able to note their visit and reason for visit, the patient met with an healthcare professional, etc)

SUMMARY:
The mobile health clinic evaluation study examines the impact of mobile health clinics on access reproductive and sexual healthcare services in underserved communities. Multiple mobile clinics operating throughout the U.S. are participating by implementing the same evaluation plan for their programs and contributing de-identified data into a shared database. This allows the investigators to both determine the impact of individual programs and to compare and contrast their impact across different programs, states, population densities (rural, urban, suburban), and populations.

DETAILED DESCRIPTION:
The purpose of this prospective/retrospective cohort study is to evaluate the effectiveness of each individual participating mobile health clinic in improving their community's health and access to care, and to compare each clinic's performance and reach within their respective communities. This Institutional Review Board (IRB)-exempt study is a descriptive review of de-identified evaluation, clinical, and operations data, including staff and patient surveys, patient metrics, and clinic operations metrics. The investigators anticipate that additional mobile clinic programs will submit de-identified data from evaluations done under local IRB exemption. The study will utilize data already collected or to be collected by each mobile health clinic as a part of its clinical and operational activities. Each mobile health clinic will decide which indicators from the evaluation instrument it will use for its own evaluation, and which will be reported to the shared database, depending on the specific services provided and population served. Data will be tracked on a per-patient-visit level or per-operational day, whichever is more relevant to the variable at hand. Data will be sourced from each mobile health clinic's current evaluation sources, including patient intake records (for demographic information, clinic visit dates, clinic procedures done), time and budget tracking software (for hours/patient and cost/patient spent), patient questionnaires (for patient satisfaction and attitudes about their mobile health clinic visit), patient post-visit follow-up questionnaires (for simple referral or prescription follow-up), and clinic operational records (for distance traveled).

ELIGIBILITY:
Inclusion Criteria:

* Patient at a participating mobile clinic

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient data included in the study will be from those who:
  1. Presented to mobile health clinic during the study periods AND,
  2. Completed an interaction with the mobile health clinic during the study periods, on which adequate evaluative data was collected on the patient visit (e.g. staff was able to note their visit and reason for visit, the patient met with a healthcare professional, etc)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Sexual Health | 1 Day
  Completed if patient received human immunodeficiency virus (HIV) status, HIV testing, education, and/or Pre-exposure prophylaxis (PrEP) AND/OR if patient received Sexually transmitted disease (STD) status, STD testing, education, and/or medication.
Vaccinations | 1 Day
  Completed if patient received human papilloma virus (HPV) vaccine or if HPV vaccination status was recorded AND/OR if the patient received any other routine, non-COVID-19 vaccine(s).
Reproductive Health | 1 Day
  Completed if patient received a pregnancy test AND/OR reported patient pregnancy status and history, prior pregnancy information, and provision of pregnancy and related referrals by the Mobile Health Clinic AND/OR if the patient received a pap smear during the visit or provided their pap smear history AND/OR if the mobile health clinic offered and provided contraception counseling and collected patient's current contraception status and contraception history AND/OR if patient requested for specific contraception or change in method AND/OR if patient received condoms AND/OR if patient received emergency contraception.
Patient screening and referrals | 1 Day
  Completed if mobile health clinic collected patient's self-reported level of health AND/OR if the patient received primary care screenings (Chol, BP, Blood sugar, A1C) AND/OR if the patient was screened for sexual assault, depression, domestic violence, and drug use, AND/OR if the patient received referrals for social services, additional health services (including specialty services), AND/OR financial or health insurance-related assistance AND/OR if the patient attended ther referral appointment AND/OR if the patient received any prescription(s) for medication, AND/OR if the mobile health clinic registered the patient to vote, AND/OR if the patient used any of the telehealth hotspot to connect with alternate providers AND/OR if the mobile health clinic staff supported the telehealth visit.
Coronavirus Disease 2019 (COVID-19) | 1 Day
  Completed if the mobile health clinic collected the patient's history on COVID-19 testing and history of COVID-19 AND/OR if the patient has been able to access COVID-19 testing AND/OR if the patient has been able to access the COVID-19 vaccination(s) and their vaccination status.

SECONDARY OUTCOMES:
Patient Demographics | 1 Day
  Completed if mobile health clinic collected data on patient's gender, transgender identity, age, sexual orientation, ethnic or racial group, highest attained education, current employment status, marital status, and new patient status.
Patient Visit | 1 Day
  Completed if mobile health clinic collected information on date of patient visit, time of arrival, time of departure, how the patient travelled to the mobile health clinic (e.g. walk, drive, public transport), how patient learned about the mobile health clinic, the approximate distance from the mobile health clinic (in miles), whether the mobile health clinic or the brick and mortar site was preferred, the mobile health clinic location at time of visit, whether the appointment was through telehealth or in- person, the patient's main reason for the visit, the type of care provided, the services that the patient wanted but could not receive, the patient's health insurance type (private, public etc.), and the cost of services provided.
Patients Assets, Risks, and Experiences | 1 Day
  Completed if the mobile health clinic collected information on patient's family size, patient's approximate income bracket and %federal poverty level (FPL), whether the patient has been able to access basic and necessary goods (e.g., food, clothing, etc.), whether the patient has been able to maintain a healthy diet, the patient's history of any chronic disease (e.g., obesity, diabetes, high BP). Whether the patient has access to transportation, healthcare services, and/or medications, if the patient has delayed services, the patient's current housing situation, the patient's history of incarceration or criminal proceedings, the patient's psychosocial circumstances related to partner or living situation, and the patient's veteran status.
Patient Satisfaction on Visit | 1 Day
  Information on how the patient heard about the clinic, patient satisfaction on a Likert scale including reason(s) for dissatisfaction (if any), any services that were wanted but not provided, the patient's likelihood to refer the clinic to others, and the patient's alternative sources of care (e.g., regular doctor, hospital/ER, urgent care).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Florida Mobile Outreach Clinic, Gainesville, Florida
  - Just the Pill, Saint Paul, Minnesota
  - Plan A Health, Inc, Louise, Mississippi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi H, Steptoe A, Heisler M, Clarke P, Schoeni RF, Jivraj S, Cho TC, Langa KM. Comparison of Health Outcomes Among High- and Low-Income Adults Aged 55 to 64 Years in the US vs England. JAMA Intern Med. 2020 Sep 1;180(9):1185-1193. doi: 10.1001/jamainternmed.2020.2802. PMID 32897385
- [Background] Rosenblatt RA, Hart LG. Physicians and rural America. West J Med. 2000 Nov;173(5):348-51. doi: 10.1136/ewjm.173.5.348. No abstract available. PMID 11069878
- [Background] Hill CF, Powers BW, Jain SH, Bennet J, Vavasis A, Oriol NE. Mobile health clinics in the era of reform. Am J Manag Care. 2014 Mar;20(3):261-4. PMID 24884754
- [Background] Yu SWY, Hill C, Ricks ML, Bennet J, Oriol NE. The scope and impact of mobile health clinics in the United States: a literature review. Int J Equity Health. 2017 Oct 5;16(1):178. doi: 10.1186/s12939-017-0671-2. PMID 28982362
- See also: National Healthcare Quality and Disparities Report — http://www.ahrq.gov/research/findings/nhqrdr/nhqdr19/index.html
- See also: Mobile Clinic Delivers Culturally Competent Services to Underserved Neighborhoods, Leading to Identification of Untreated Chronic Conditions, Better Blood Pressure Control, and Significant Return on Investment | AHRQ Health Care Innovations Exchange — https://innovations.ahrq.gov/profiles/mobile-clinic-delivers-culturally-competent-services-underserved-neighborhoods-leading#1